CLINICAL TRIAL: NCT06327607
Title: Psychosexuological Interventions to Support Sexual Function in Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1952
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Standard iter of treatment for breast cancer
  Interventions: Other: Control Group
- Experimental group: Psychosexuological intervention
  Interventions: Other: Psychosexological intervention

INTERVENTIONS:
Other: Control Group — Standard care for breast cancer
  Groups: Control group
Other: Psychosexological intervention — The intervention will be conducted individually and will take place once a week for one hour, for a total of 8 consecutive weeks, which must be completed within a maximum duration of 10 weeks.
  Groups: Experimental group

SUMMARY:
Prospective pilot study on the feasibility and efficacy of a brief psychosexual support intervention in breast cancer patients undergoing hormonal therapies for at least 6 months.

The study is randomized in the two following arms:

Control arm (standard care pathway) Psychosexual intervention arm

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effectiveness of a psychosexual intervention on sexual functioning, mood (levels of depression and anxiety), sleep, and quality of life, compared to standard care pathway. Considering the high incidence of sexual dysfunction in breast cancer patients, this study will focus on this population of patients.

The psychosexual intervention aims to improve female sexual functionality and satisfaction by facilitating the understanding of disorders, enabling adequate assessment of possible interventions, and adopting specific treatment exercises.

Patients will be randomized in one of the following two arms:

Control arm (standard care pathway) Psychosexual intervention arm

ELIGIBILITY:
Inclusion Criteria:

* Women with age >=18 years;
* Breast cancer patients undergoing hormonal therapy for at least 6 months in accordance with clinical practice and scientific evidence;
* Pre-menopausal patients (regular menstrual cycles in the last year) before the start of oncological treatments;
* Presence of one or more criteria of sexual dysfunction as per DSM-5;
* Acceptance and signature of the Informed Consent.

Exclusion Criteria:

* Patients in postmenopausal status;
* Presence of psychiatric or neurological conditions that impair the ability to perform the exercises proposed by the research project;
* Already undergoing psycho-sexual counseling;
* Refusal to sign the informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is for women who have had breast cancer and are currently undergoing hormonal therapies.
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of differences between two arms in female sexual satisfaction and functionality scores | 10 weeks
  Measurement of the differences between the two groups in female sexual satisfaction and functionality scores before and after participation in the psychosexual intervention group, we will use the Brief Index of Sexual Functioning-Woman (BISF-W). This is a self-administered questionnaire specifically designed to assess female sexual functionality and satisfaction.

SECONDARY OUTCOMES:
Evaluation of differences between two arms in levels of quality of life | 10 weeks
  To measure the differences between the two arms in levels of quality of life investigated using the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire.
Evaluation of differences between two arms in levels of anxiety and depression | 10 weeks
  Levels of anxiety and depression measured using the Hospital Anxiety and Depression Scale (HADS).
Evaluation of differences between two arms in levels of sleep quality | 10 weeks
  Levels of sleep quality measured using the Pittsburgh Sleep Quality Index (PSQI) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Pravettoni, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy